CLINICAL TRIAL: NCT00859703
Title: Randomized, Double-blinded, Placebo Controlled Study to Assess Efficacy of Oral 35 mg Per Week Risedronate in Preventing Bone Loss in Postmenopausal Women With Aromatase Inhibitor Therapy for Breast Cancer.
Brief Title: Study to Assess Efficacy of Risedronate in Preventing Bone Loss in Postmenopausal Women Treated for Breast Cancer
Acronym: RISAROS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006.45346
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Breast Cancer; Menopause; Osteopenia
Keywords: Aromatase inhibitor treatment; osteoporosis; breast cancer; bisphosphonates
MeSH Terms: conditions — Breast Neoplasms; Bone Diseases, Metabolic; Osteoporosis | interventions — Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator): Patients receive placebo 35 mg once a week plus a calcium and vitamin D supplementation.
  Measure of bone density, bone markers, clinical examination and questionnaire regarding fractures will be assessed at 12 and 24 months of treatment
  Interventions: Drug: Placebo
- 1 (Active Comparator): Patients receive risedronate 35 mg once a week plus a calcium and vitamin D supplementation.
  Measure of bone density, bone markers, clinical examination and questionnaire regarding fractures will be assessed at 12 and 24 months of treatment
  Interventions: Drug: Risedronate

INTERVENTIONS:
Drug: Risedronate — 35mg oral risedronate once per week for 24 months
  Arms: 1
Drug: Placebo — Placebo 35 mg once a week for 24 months
  Arms: 2

SUMMARY:
Aromatase inhibitor therapy is in France the adjuvant reference treatment for postmenopausal women with early-stage breast cancer. This treatment induces bone loss and a higher risk of fractures.

This study aimed to document the effect of bisphosphonate therapy in preventing bone loss and osteoporotic fractures in postmenopausal women with aromatase inhibitor treatment for breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (more than one year since last menstrual period or removal of ovarian function by surgical or radiotherapic means)
* Operated for an invasive breast cancer (histologically proven)
* Surgical treatment completed and cycles of adjuvant chemotherapy (if necessary) completed
* Treated with aromatase inhibitor
* Osteopenic (-2.5<T score<-1) without osteoporotic fracture
* With written informed consent signed
* With social security

Exclusion Criteria:

* Women presenting a history of osteoporotic fracture or a T score less than -2.5 at at least one measure site
* Women presenting clinical signs of metastases
* Having received other hormonal treatment in the last 3 months
* Having received treatment by bisphosphonates, raloxifene, tamoxifen, parathormone, strontium ranelate, tibolone,calcitonin and corticosteroids at more than 5mg/d for 3 months in the last year
* Presenting a known and untreated hyperthyroid
* Presenting a known hyperadrenocorticism
* Patients treated and followed for Paget's disease of bone
* Presenting a untreated primary hyperparathyroid
* Presenting an indication against risedronate (known hypersensibility to risedronate monosodium and/or one of its excipients, non-corrected hypocalcemia, pregnancy or breast feeding, severe renal insufficiency inferior to 30 ml/min)
* Patients presenting malabsorption syndrome for glucose/galactose
* Person participating in another clinical trial concerning a medicine susceptible to influence bone mass

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Evolution of the lumbar spine Bone Mineral Density after one year of treatment | 1 year

SECONDARY OUTCOMES:
Evolution of femoral BMD after one year of treatment | 1 year
Evolution of lumbar spine and femoral BMD after two years of treatment | 2 years
Evolution of bone resorption and formation markers | 2 years
Proportion of fractures after two years of treatment | 2 years
Evolution of estradiol levels | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie Fontana, M.D, Principal Investigator — Hôpital Edouard Herriot
Locations (1):
- Service de Rhumatology et de Pathologie Osseuse, Hôpital Edouard Herriot, Lyon, France

REFERENCES:
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716